CLINICAL TRIAL: NCT04829890
Title: Adjuvant Dose-dense Sequential Chemotherapy With Epirubicin, CMF, and Weekly Docetaxel or Weekly Paclitaxel in Patients With Resected High-risk Breast Cancer: A Hellenic Cooperative Oncology Group (HeCOG) Study
Brief Title: Adjuvant Chemotherapy With Epirubicin, CMF, and Weekly Docetaxel or Weekly Paclitaxel in Patients With Resected High-risk Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: HE10/04
Record Dates: First submitted 2021-03-29; First posted 2021-04-02 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer; Adenocarcinoma of Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was a transnational pooled analysis of biological material from patients with resected high risk breast cancer who had received adjuvant chemotherapy with epirubicin and cyclophosphamide followed by weekly docetaxel or weekly paclitaxel.

DETAILED DESCRIPTION:
This was a transnational analysis of biological material from patients with resected high risk breast cancer who are treated at Hellenic Cooperative Oncology Group (HeCOG) affiliated departments of oncology. This study was a pooled analysis of two separate sequential feasibility studies who received the below described treatment. Patients who participated were 18 years old or older, women of any menopausal status who received epirubicin for 3 cycles every 2 weeks followed by 3 cycles with cyclophosphamide every 2 weeks followed 3 weeks later by 9 weekly cycles with docetaxel or paclitaxel. G-CSF was given on days 2-7 of each cycle during treatment with Epirubicin and cyclophosphamide. All premenopausal patients with receptor positive status received tamoxifen 20 mg p.o. daily for 5 years. All postmenopausal patients with receptor positive status were treated with anastrazole 1mg for 5 years. RT was required for all patients (pre- or post -menopausal), providing that they had either a partial mastectomy or tumor size > 5cm and /or more than 4 positive lymph nodes, irrespectively the type of surgery (conservative or radical).

ELIGIBILITY:
Inclusion Criteria:

* Histology-confirmed epithelial cancer of the mammary gland.
* Pre and post menopausal patients with early breast cancer and involved axillary lymph nodes (T 1-3 N1 M0) or high-risk N0 patients. A N0 patient is considered "high-risk" if she fulfills at least one of the following criteria; T>= 2cm, Estrogen Receptor (ER)/Progesterone receptor (PgR) negative, HER-2 3+, infiltration of blood or lymphatic vessels or nerves, grade 3.
* White Blood Cell count (WBC) > 4 x 109 / l, platelets > 100 x 109 / l.
* Serum creatinine, Aspartate aminotransferase (AST/SGOT),Alanine aminotransferase (ALT/SGPT), gamma-glutamyltransferase, serum bilirubin 1.3 mg/ml inside the normal range of the participating hospital.
* Performance status (WHO) 0 or 1.
* Age >=18 years
* Previous surgical treatment: Either radical surgery or, for a partial mastectomy, a histologically confirmed safe margin of 2 cm or more and the results of the axillary node dissection available.
* No evidence of significant cardiac disease

Exclusion Criteria:

* History of myocardial infarction within the previous 12 months or heart failure (including cardiac insufficiency controlled by digitalis and diuretics) or arrhythmias requiring medication or uncontrolled arterial hypertension (BP> 200/110 mm Hg). A normal baseline Left Ventricular Ejection Fraction (LVEF) should be demonstrated by multigated acquisition (MUGA) scan or echocardiogram.
* No previous antitumor chemotherapy or radiation
* Time from surgery 2 to 4 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This is a transnational pooled analysis, feasibility study from two sequential studies with biological material from patients with confirmed breast cancer with high risk of recurrence. Patients have been treated in Hellenic Cooperative Oncology Group (HeCOG) affiliated departments of oncology.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2004-02 (Actual); Primary Completion 2006-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Evaluating the feasibility profile of dose dense sequential chemotherapy with Epirubicin, cyclophosphamide and weekly docetaxel or weekly paclitaxel. | Up to 147 days
Number of Participants with Treatment-Related Adverse Events treated with dose dense sequential chemotherapy with Epirubicin, cyclophosphamide and weekly docetaxel or weekly paclitaxel. | Up to 147 days

REFERENCES:
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG). Effects of chemotherapy and hormonal therapy for early breast cancer on recurrence and 15-year survival: an overview of the randomised trials. Lancet. 2005 May 14-20;365(9472):1687-717. doi: 10.1016/S0140-6736(05)66544-0. PMID 15894097
- [Background] Norton L. Theoretical concepts and the emerging role of taxanes in adjuvant therapy. Oncologist. 2001;6 Suppl 3:30-5. doi: 10.1634/theoncologist.6-suppl_3-30. PMID 11346683
- [Background] Citron ML. Dose density in adjuvant chemotherapy for breast cancer. Cancer Invest. 2004;22(4):555-68. doi: 10.1081/cnv-200027134. PMID 15565814
- [Background] Colozza M, de Azambuja E, Cardoso F, Bernard C, Piccart MJ. Breast cancer: achievements in adjuvant systemic therapies in the pre-genomic era. Oncologist. 2006 Feb;11(2):111-25. doi: 10.1634/theoncologist.11-2-111. PMID 16476832
- [Background] Henderson IC, Berry DA, Demetri GD, Cirrincione CT, Goldstein LJ, Martino S, Ingle JN, Cooper MR, Hayes DF, Tkaczuk KH, Fleming G, Holland JF, Duggan DB, Carpenter JT, Frei E 3rd, Schilsky RL, Wood WC, Muss HB, Norton L. Improved outcomes from adding sequential Paclitaxel but not from escalating Doxorubicin dose in an adjuvant chemotherapy regimen for patients with node-positive primary breast cancer. J Clin Oncol. 2003 Mar 15;21(6):976-83. doi: 10.1200/JCO.2003.02.063. PMID 12637460
- [Background] Hudis, C.; Citron, M.; Berry, D.; Cirrincione, C.; Gradishar, W.; Davidson, N.; Martino, S.; Livingston, R.; Ingle, J.; Perez, E.; Abrams, J.; Schilsky, R.; Ellis, M.; Muss, H.; Norton, L.; Winer E. Five year follow-up of INT C9741: dose-dense (DD) chemotherapy (CRx) is safe and effective. San Antonio Breast Cancer Symposium 2005, Abstract 41
- [Background] Mamounas EP, Bryant J, Lembersky B, Fehrenbacher L, Sedlacek SM, Fisher B, Wickerham DL, Yothers G, Soran A, Wolmark N. Paclitaxel after doxorubicin plus cyclophosphamide as adjuvant chemotherapy for node-positive breast cancer: results from NSABP B-28. J Clin Oncol. 2005 Jun 1;23(16):3686-96. doi: 10.1200/JCO.2005.10.517. Epub 2005 May 16. PMID 15897552
- [Background] Crown, J.P.; Francis, P.; Di Leo, A.; Buyse, M.; Balil, A.; Anderson, M.; Nordenskj¨ old, B.; Jakesz, R.; Gutierrez J.; PiccartM. Docetaxel (T) given concurrently with or sequentially to anthracycline-based (A) adjuvant therapy (adjRx) for patients (pts) with node-positive (N+) breast cancer (BrCa), in comparison with non-T adjRx: First results of the BIG 2-98 Trial at 5 years median follow-up (MFU). J Clin Oncol, 2006 ASCO Annual Meeting Proceedings Part I. Vol 24, No. 18S (June 20 Supplement), 2006: LBA519
- [Background] Fountzilas G, Skarlos D, Dafni U, Gogas H, Briasoulis E, Pectasides D, Papadimitriou C, Markopoulos C, Polychronis A, Kalofonos HP, Siafaka V, Kosmidis P, Timotheadou E, Tsavdaridis D, Bafaloukos D, Papakostas P, Razis E, Makrantonakis P, Aravantinos G, Christodoulou C, Dimopoulos AM. Postoperative dose-dense sequential chemotherapy with epirubicin, followed by CMF with or without paclitaxel, in patients with high-risk operable breast cancer: a randomized phase III study conducted by the Hellenic Cooperative Oncology Group. Ann Oncol. 2005 Nov;16(11):1762-71. doi: 10.1093/annonc/mdi366. Epub 2005 Sep 7. PMID 16148021
- [Background] Eniu A, Palmieri FM, Perez EA. Weekly administration of docetaxel and paclitaxel in metastatic or advanced breast cancer. Oncologist. 2005 Oct;10(9):665-85. doi: 10.1634/theoncologist.10-9-665. PMID 16249346
- [Background] Seidman AD, Hudis CA, Albanell J, Tong W, Tepler I, Currie V, Moynahan ME, Theodoulou M, Gollub M, Baselga J, Norton L. Dose-dense therapy with weekly 1-hour paclitaxel infusions in the treatment of metastatic breast cancer. J Clin Oncol. 1998 Oct;16(10):3353-61. doi: 10.1200/JCO.1998.16.10.3353. PMID 9779712
- [Background] Wist EA, Sommer HH, Ostenstad B, Risberg T, Fjaestad K. Weekly one-hour paclitaxel as first-line chemotherapy for metastatic breast cancer. Acta Oncol. 2004;43(1):11-4. doi: 10.1080/02841860310017748. PMID 15068314
- [Background] Sato K, Inoue K, Saito T, Kai T, Mihara H, Okubo K, Koh J, Mochizuki H, Tabei T; Saitama Breast Cancer Clinical Study Group. Multicenter phase II trial of weekly paclitaxel for advanced or metastatic breast cancer: the Saitama Breast Cancer Clinical Study Group (SBCCSG-01). Jpn J Clin Oncol. 2003 Aug;33(8):371-6. doi: 10.1093/jjco/hyg075. PMID 14523055
- [Background] Gori S, Mosconi AM, Basurtol C, Cherubinil R, De Angelis V, Tonato M, Colozza M. Weekly paclitaxel in metastatic breast cancer patients: a phase II study. Tumori. 2002 Nov-Dec;88(6):470-3. doi: 10.1177/030089160208800607. PMID 12597140
- [Background] Perez EA, Vogel CL, Irwin DH, Kirshner JJ, Patel R. Multicenter phase II trial of weekly paclitaxel in women with metastatic breast cancer. J Clin Oncol. 2001 Nov 15;19(22):4216-23. doi: 10.1200/JCO.2001.19.22.4216. PMID 11709565
- [Background] Perez EA, Vogel CL, Irwin DH, Kirshner JJ, Patel R. Weekly paclitaxel in women age 65 and above with metastatic breast cancer. Breast Cancer Res Treat. 2002 May;73(1):85-8. doi: 10.1023/a:1015230212550. PMID 12083634
- [Background] Seidman, A.D.; Berry, D.; Cirrincione, C.; Harris, L.; Dressler, L.; Muss, H.; Naughton, M.; Norton, L.; Winer, E.; Hudis, C. CALGB 9840: Phase III study of weekly (W) paclitaxel (P) via 1-hour (h) infusion versus standard (S) 3h infusion every third week in the treatment of metastatic breast cancer (MBC), with trastuzumab(T) for HER2 positive MBC and randomized for T in HER2 normal MBC. J Clin Oncol 2004, 22 (Suppl), 14S (abstract 512).
- [Background] Sparano, J.A.; Wang, M.; Martino, S.; Jones, V.; Perez, E.A.; Saphner, T.; Wolff, A.C.; Sledge, G.W.; Wood, W.C.; Davidson, N.E. Phase III study of doxorubicin-cyclophosphamide followed by paclitaxel or docetaxel given every 3 weeks or weekly in patients with axillary node-positive or high-risk node-negative breast cancer: results of North American Breast Cancer Intergroup Trial E1199. 28th Annual San Antonio Breast Cancer Symposium 2005.Breast Cancer Res Treat 2005, 94 (Suppl 1) (abstract 48).
- [Background] Fountzilas G, Pectasides D, Christodoulou C, Timotheadou E, Economopoulos T, Papakostas P, Papadimitriou C, Gogas H, Efstratiou I, Skarlos D. Adjuvant dose-dense sequential chemotherapy with epirubicin, CMF, and weekly docetaxel is feasible and safe in patients with operable breast cancer. Med Oncol. 2006;23(4):479-88. doi: 10.1385/MO:23:4:479. PMID 17303906
- [Background] Goldhirsch A, Glick JH, Gelber RD, Coates AS, Thurlimann B, Senn HJ; Panel members. Meeting highlights: international expert consensus on the primary therapy of early breast cancer 2005. Ann Oncol. 2005 Oct;16(10):1569-83. doi: 10.1093/annonc/mdi326. Epub 2005 Sep 7. PMID 16148022
- [Background] Hryniuk W, Levine MN. Analysis of dose intensity for adjuvant chemotherapy trials in stage II breast cancer. J Clin Oncol. 1986 Aug;4(8):1162-70. doi: 10.1200/JCO.1986.4.8.1162. PMID 3525765
- [Background] Hryniuk WM, Levine MN, Levin L. Analysis of dose intensity for chemotherapy in early (stage II) and advanced breast cancer. NCI Monogr. 1986;(1):87-94. PMID 3534595
- [Background] Von Hoff DD, Clark GM, Weiss GR, Marshall MH, Buchok JB, Knight WA 3rd, LeMaistre CF. Use of in vitro dose response effects to select antineoplastics for high-dose or regional administration regimens. J Clin Oncol. 1986 Dec;4(12):1827-34. doi: 10.1200/JCO.1986.4.12.1827. PMID 2431110
- [Background] Fisher B, Anderson S, Wickerham DL, DeCillis A, Dimitrov N, Mamounas E, Wolmark N, Pugh R, Atkins JN, Meyers FJ, Abramson N, Wolter J, Bornstein RS, Levy L, Romond EH, Caggiano V, Grimaldi M, Jochimsen P, Deckers P. Increased intensification and total dose of cyclophosphamide in a doxorubicin-cyclophosphamide regimen for the treatment of primary breast cancer: findings from National Surgical Adjuvant Breast and Bowel Project B-22. J Clin Oncol. 1997 May;15(5):1858-69. doi: 10.1200/JCO.1997.15.5.1858. PMID 9164196
- [Background] Fisher B, Anderson S, DeCillis A, Dimitrov N, Atkins JN, Fehrenbacher L, Henry PH, Romond EH, Lanier KS, Davila E, Kardinal CG, Laufman L, Pierce HI, Abramson N, Keller AM, Hamm JT, Wickerham DL, Begovic M, Tan-Chiu E, Tian W, Wolmark N. Further evaluation of intensified and increased total dose of cyclophosphamide for the treatment of primary breast cancer: findings from National Surgical Adjuvant Breast and Bowel Project B-25. J Clin Oncol. 1999 Nov;17(11):3374-88. doi: 10.1200/JCO.1999.17.11.3374. PMID 10550131
- [Background] French Adjuvant Study Group. Benefit of a high-dose epirubicin regimen in adjuvant chemotherapy for node-positive breast cancer patients with poor prognostic factors: 5-year follow-up results of French Adjuvant Study Group 05 randomized trial. J Clin Oncol. 2001 Feb 1;19(3):602-11. doi: 10.1200/JCO.2001.19.3.602. PMID 11157009
- [Background] Fornier MN, Seidman AD, Lake D, D'Andrea G, Bromberg J, Robson M, Van Poznak C, Panageas KS, Atienza M, Norton L, Hudis C. Increased dose density is feasible: a pilot study of adjuvant epirubicin and cyclophosphamide followed by paclitaxel, at 10- or 11-day intervals with filgrastim support in women with breast cancer. Clin Cancer Res. 2007 Jan 1;13(1):223-7. doi: 10.1158/1078-0432.CCR-06-1731. PMID 17200358
- [Background] Dang CT, D'Andrea GM, Moynahan ME, Dickler MN, Seidman AD, Fornier M, Robson ME, Theodoulou M, Lake D, Currie VE, Hurria A, Panageas KS, Norton L, Hudis CA. Phase II study of feasibility of dose-dense FEC followed by alternating weekly taxanes in high-risk, four or more node-positive breast cancer. Clin Cancer Res. 2004 Sep 1;10(17):5754-61. doi: 10.1158/1078-0432.CCR-04-0634. PMID 15355903
- [Background] Tabernero J, Climent MA, Lluch A, Albanell J, Vermorken JB, Barnadas A, Anton A, Laurent C, Mayordomo JI, Estaun N, Losa I, Guillem V, Garcia-Conde J, Tisaire JL, Baselga J. A multicentre, randomised phase II study of weekly or 3-weekly docetaxel in patients with metastatic breast cancer. Ann Oncol. 2004 Sep;15(9):1358-65. doi: 10.1093/annonc/mdh349. PMID 15319242
- [Background] Crown J, O'Leary M, Ooi WS. Docetaxel and paclitaxel in the treatment of breast cancer: a review of clinical experience. Oncologist. 2004;9 Suppl 2:24-32. doi: 10.1634/theoncologist.9-suppl_2-24. PMID 15161988
- [Background] Esteva FJ, Valero V, Booser D, Guerra LT, Murray JL, Pusztai L, Cristofanilli M, Arun B, Esmaeli B, Fritsche HA, Sneige N, Smith TL, Hortobagyi GN. Phase II study of weekly docetaxel and trastuzumab for patients with HER-2-overexpressing metastatic breast cancer. J Clin Oncol. 2002 Apr 1;20(7):1800-8. doi: 10.1200/JCO.2002.07.058. PMID 11919237
- [Background] Anan K, Mitsuyama S, Taniguchi H, Yamamoto Y, Fujiyoshi K, Tateishi T, Tamura K. [Adjuvant doxorubicin and cyclophosphamide followed by weekly paclitaxel for Japanese women with node-positive breast cancer: a multi-institutional feasibility study in a variety of practice settings in Kyushu]. Gan To Kagaku Ryoho. 2006 Oct;33(10):1417-22. Japanese. PMID 17033230
- [Background] Green MC, Buzdar AU, Smith T, Ibrahim NK, Valero V, Rosales MF, Cristofanilli M, Booser DJ, Pusztai L, Rivera E, Theriault RL, Carter C, Frye D, Hunt KK, Symmans WF, Strom EA, Sahin AA, Sikov W, Hortobagyi GN. Weekly paclitaxel improves pathologic complete remission in operable breast cancer when compared with paclitaxel once every 3 weeks. J Clin Oncol. 2005 Sep 1;23(25):5983-92. doi: 10.1200/JCO.2005.06.232. Epub 2005 Aug 8. PMID 16087943
- [Background] Ellis GK, Barlow WE, Gralow JR, Hortobagyi GN, Russell CA, Royce ME, Perez EA, Lew D, Livingston RB. Phase III comparison of standard doxorubicin and cyclophosphamide versus weekly doxorubicin and daily oral cyclophosphamide plus granulocyte colony-stimulating factor as neoadjuvant therapy for inflammatory and locally advanced breast cancer: SWOG 0012. J Clin Oncol. 2011 Mar 10;29(8):1014-21. doi: 10.1200/JCO.2009.27.6543. Epub 2011 Jan 10. PMID 21220618
- [Background] Citron ML, Berry DA, Cirrincione C, Hudis C, Winer EP, Gradishar WJ, Davidson NE, Martino S, Livingston R, Ingle JN, Perez EA, Carpenter J, Hurd D, Holland JF, Smith BL, Sartor CI, Leung EH, Abrams J, Schilsky RL, Muss HB, Norton L. Randomized trial of dose-dense versus conventionally scheduled and sequential versus concurrent combination chemotherapy as postoperative adjuvant treatment of node-positive primary breast cancer: first report of Intergroup Trial C9741/Cancer and Leukemia Group B Trial 9741. J Clin Oncol. 2003 Apr 15;21(8):1431-9. doi: 10.1200/JCO.2003.09.081. Epub 2003 Feb 13. PMID 12668651
- [Background] Martin M, Pienkowski T, Mackey J, Pawlicki M, Guastalla JP, Weaver C, Tomiak E, Al-Tweigeri T, Chap L, Juhos E, Guevin R, Howell A, Fornander T, Hainsworth J, Coleman R, Vinholes J, Modiano M, Pinter T, Tang SC, Colwell B, Prady C, Provencher L, Walde D, Rodriguez-Lescure A, Hugh J, Loret C, Rupin M, Blitz S, Jacobs P, Murawsky M, Riva A, Vogel C; Breast Cancer International Research Group 001 Investigators. Adjuvant docetaxel for node-positive breast cancer. N Engl J Med. 2005 Jun 2;352(22):2302-13. doi: 10.1056/NEJMoa043681. PMID 15930421
- [Background] Sparano JA, et al. Phase III study of doxorubicin-cyclophosphamide followed by paclitaxel or docetaxel given every 3 weeks or weekly in patients with axillary node-positive or high-risk node-negative breast cancer: results of North American Breast Cancer Intergroup Trial E1199. (Abstr 48) 28th Annual San Antonio Breast Cancer Symposium 2005. Breast Cancer Res Treat 2005; 94 (Suppl 1).
- [Background] Chan S, Friedrichs K, Noel D, Pinter T, Van Belle S, Vorobiof D, Duarte R, Gil Gil M, Bodrogi I, Murray E, Yelle L, von Minckwitz G, Korec S, Simmonds P, Buzzi F, Gonzalez Mancha R, Richardson G, Walpole E, Ronzoni M, Murawsky M, Alakl M, Riva A, Crown J; 303 Study Group. Prospective randomized trial of docetaxel versus doxorubicin in patients with metastatic breast cancer. J Clin Oncol. 1999 Aug;17(8):2341-54. doi: 10.1200/JCO.1999.17.8.2341. PMID 10561296
- [Background] Jones SE, Erban J, Overmoyer B, Budd GT, Hutchins L, Lower E, Laufman L, Sundaram S, Urba WJ, Pritchard KI, Mennel R, Richards D, Olsen S, Meyers ML, Ravdin PM. Randomized phase III study of docetaxel compared with paclitaxel in metastatic breast cancer. J Clin Oncol. 2005 Aug 20;23(24):5542-51. doi: 10.1200/JCO.2005.02.027. PMID 16110015
- [Background] Hainsworth JD, Burris HA 3rd, Erland JB, Thomas M, Greco FA. Phase I trial of docetaxel administered by weekly infusion in patients with advanced refractory cancer. J Clin Oncol. 1998 Jun;16(6):2164-8. doi: 10.1200/JCO.1998.16.6.2164. PMID 9626217
- [Background] Briasoulis E, Karavasilis V, Anastasopoulos D, Tzamakou E, Fountzilas G, Rammou D, Kostadima V, Pavlidis N. Weekly docetaxel in minimally pretreated cancer patients: a dose-escalation study focused on feasibility and cumulative toxicity of long-term administration. Ann Oncol. 1999 Jun;10(6):701-6. doi: 10.1023/a:1008399712913. PMID 10442193
- [Background] Burstein HJ, Manola J, Younger J, Parker LM, Bunnell CA, Scheib R, Matulonis UA, Garber JE, Clarke KD, Shulman LN, Winer EP. Docetaxel administered on a weekly basis for metastatic breast cancer. J Clin Oncol. 2000 Mar;18(6):1212-9. doi: 10.1200/JCO.2000.18.6.1212. PMID 10715290
- [Background] Stemmler J, Mair W, Stauch M, Papke J, Deutsch G, Abenhardt W, Dorn B, Kentenich C, Malekmohammadi M, Jackisch C, Leinung S, Brudler O, Vehling-Kaiser U, Stamp J, Heinemann V. High efficacy and low toxicity of weekly docetaxel given as first-line treatment for metastatic breast cancer. Oncology. 2005;68(1):71-8. doi: 10.1159/000084823. Epub 2005 Mar 12. PMID 15809523
- [Background] Di Leo A, Crown J, Nogaret JM, Duffy K, Bartholomeus S, Dolci S, Rowan S, O'Higgins N, Paesmans M, Larsimont D, Riva A, Piccart MJ. A feasibility study evaluating docetaxel-based sequential and combination regimens in the adjuvant therapy of node-positive breast cancer. Ann Oncol. 2000 Feb;11(2):169-75. doi: 10.1023/a:1008345432342. PMID 10761751
- [Background] Fumoleau P, et al. Adjuvant dose-dense (3 FEC 100 followed 3 docetaxel every 2 weeks) regimen is not feasible. Results of the FNCLCC-PACS 06 Study. (Abstr 2071) 28th Annual San Antonio Breast Cancer Symposium 2005.Breast Cancer Res Treat 2005; 94(Suppl 1): S108
- [Background] Miller KD, McCaskill-Stevens W, Sisk J, Loesch DM, Monaco F, Seshadri R, Sledge GW Jr. Combination versus sequential doxorubicin and docetaxel as primary chemotherapy for breast cancer: A randomized pilot trial of the Hoosier Oncology Group. J Clin Oncol. 1999 Oct;17(10):3033-7. doi: 10.1200/JCO.1999.17.10.3033. PMID 10506597
- [Background] Miller KD, Soule SE, Calley C, Emerson RE, Hutchins GD, Kopecky K, Badve S, Storniolo A, Goulet R, Sledge GW Jr. Randomized phase II trial of the anti-angiogenic potential of doxorubicin and docetaxel; primary chemotherapy as Biomarker Discovery Laboratory. Breast Cancer Res Treat. 2005 Jan;89(2):187-97. doi: 10.1007/s10549-004-2044-y. PMID 15692762